CLINICAL TRIAL: NCT04524793
Title: Pilot Study to Investigate the Efficacy and Safety of Endovenous Microwave Ablations for Treatment of Varicose Veins in Singapore
Brief Title: Efficacy and Safety of Endovenous Microwave Ablations for Treatment of Varicose Veins in Singapore
Acronym: MAESTRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/2371
Record Dates: First submitted 2020-08-12; First posted 2020-08-24 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Venous Insufficiency; Varicose Veins; Vascular Diseases
Keywords: endovenous microwave ablation
MeSH Terms: conditions — Venous Insufficiency; Varicose Veins; Vascular Diseases | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovenous Microwave Ablations (Other): Patients that have undergone Endovenous Microwave Ablation from ECO (Nanjing ECO Microwave System Co., Ltd) to treat primary great and short saphenous vein reflux
  Interventions: Other: Questionnaires; Other: Physical examinations

INTERVENTIONS:
Other: Questionnaires — Questionnaires to assess the quality of life (EQ-5D, CVVQ, CIVIQ, AVVQ, Patient satisfaction survey)
Other: Physical examinations — GSV/SSV/AASV reflux, CEAP Classification (Clinical, Aetiological, Anatomical and Pathophysiology), Venous Clinical Severity Score (VCSS) and duplex ultrasound

SUMMARY:
The purpose of this study is to assess change in patient's symptoms before and after Endovenous Microwave Ablation (EMA) as treatment for varicose veins. At the same time, it is to evaluate the effectiveness of EMA and its treatment outcomes over a period of 1 year.

DETAILED DESCRIPTION:
Healthy leg veins have valves that allow blood to move in one direction from the lower leg to the heart. These valves open when blood is flowing toward the heart and then quickly close to stop any backward flow. When veins weaken, their valves cannot close properly, causing reversal of blood flow in the vein or venous reflux. Venous reflux due to the incompetent valves in the superficial venous system is the most common form of venous insufficiency, also known as varicose veins. This happens most often in the veins closest to the skin; the superficial veins. Varicose veins may or may not have associated symptoms and can look like twisted, bulging, rope-like cords or even small spider veins. While sometimes asymptomatic, varicose veins can be associated with pain, aching or cramping in the legs, heaviness or a tired sensation, paresthesia, pruritus, edema, inflammation with superficial phlebitis or thrombophlebitis, ulceration, bleeding from ulcerated varicosities, ecchymosis from subcutaneous rupture of varicosities, and deep venous thrombosis from extension of superficial thrombophlebitis.

Venous insufficiency of lower extremities is a very common condition that is influenced by genetic and mechanical factors, and is a chronic and progressive disorder. Prevalence estimates vary widely by geographic location, with the highest reported rates in Western countries, including Western Europe and the United States. Prevalence estimates of varicose veins range from <1% to up to 73% in females and 2% to up to 56% in males. The reported prevalence ranges presumably reflect differences in the population distribution of risk factors, accuracy in application of diagnostic criteria, and the quality and availability of medical diagnostic and treatment resources. Risk factors for venous insufficiency include older age, female gender and pregnancy, family history of venous disease, obesity and occupations associated with prolonged standing.

There are a number of treatment options available to subjects with varicose veins, including vein stripping surgery, and thermal ablation; for example, Endovenous laser ablation (EVLA), radiofrequency ablation (RFA), and sclerotherapy. Recent technological advances have also brought about new treatment methods that are non-thermal, non-tumescent (NTNT). These include Venaseal and Clarivein. The goal of each of these treatment regimens is to eliminate source of reflux in order to control the progression of the disease, improve symptoms, promote ulcer healing, and prevent recurrence or a combination of these. The latest treatment available uses microwave ablation, which is a sub-type of radiofrequency and has the same characteristics as radiofrequency ablation.

The aim of this study is to report a collaborative, prospective Singaporean experience using the ECO Varicose Veins Therapeutic Unit from ECO (Nanjing ECO Microwave System Co., Ltd) for Endovenous Microwave Ablation (EMA) to treat primary great and short saphenous vein reflux and to evaluate its safety, efficacy and performance.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years, able to understand the requirements of the study and provide informed consent.
* C2 - C5 varicose veins / CVI
* Symptomatic primary GSV, SSV or AASV incompetence, with reflux >0.5 seconds on colour duplex, including one or more of the following symptoms: aching, throbbing, heaviness, fatigue, pruritus, night cramps, restlessness, generalized pain or discomfort, swelling.
* Patients who has GSV, SSV AASV diameters of 3mm to 12mm in the standing postition.

Exclusion Criteria:

* Current DVT or history of DVT
* Recurrent varicose veins
* Pregnant patients
* Arterial disease (ABPI <0.8)
* Sepsis
* Patients who are unwilling to participate
* Inability or unwillingness to complete questionnaires
* Adverse reaction to sclerosant or cyanoacrylate
* GSV, SSV or AASV severely tortuous
* Life expectancy < 1 year
* Active treatment for malignancy other than non-melanoma skin cancer
* Current, regular use of systemic anticoagulation (e.g. warfarin, heparin)
* Daily us of narcotic analgesia or NSAIDS to control pain associated with venous disease

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Technical Success at time of procedure | Immediately post-procedure
  Occlusion of treated vein post-procedure
Anatomical Success | 2 weeks to 12 months post-procedure
  Anatomical success defined as occlusion of treated vessel, as determined by duplex ultrasound

SECONDARY OUTCOMES:
Quality of Life score using EQ-5D questionnaire | Baseline, 2-weeks, 3 months, 6 months and 12 months
  EQ-5D is used to assess quality of life based on Mobility, Self-care, Usual Activities, Pain/Discomfort and Anxiety, rated at 5 levels: no problems, slight problems, moderate problems, severe problems, unable to perform activity. Inputs from this questionnaire is used to observe for changes in quality of life overtime
Quality of life score using the Chronic Venous Insufficiency Questionnaire (CIVIQ) | Baseline, 2-weeks, 3 months, 6 months and 12 months
  CIVIQ-14 is a questionnaire based on three dimensions - pain, physical and psychological, based on a scale from 1 to 5 (no trouble, slight, moderate, considerable, severe). Based on inputs, Global Index Score (GIS) will be tabulated, ranging from 0 to 100 - the higher the value, the poorer the quality of life.
Quality of life score using the Aberdeen Varicose Veins Questionnaire (AVVQ) | Baseline, 2-weeks, 3 months, 6 months and 12 months
  To measure health status of varicose vein patients based on symptoms and impact on daily activities. A total score ranging from 0 to 100 will be tabulated, with 100 being worst quality of life
Clinical Change using Venous Clinical Severity Score (VCSS) | Baseline, 2-weeks, 3 months, 6 months and 12 months
  VCSS evaluates the severity of hallmarks of venous disease - 0 (none), 1 (Mild) , 2(Moderate), 3 (Severe).
Time taken to return to work and normal activities | 10 days post-op
  Patient will be given a diary to record the day when they return to work and normal activities.
Patient's satisfaction | 2-weeks, 3 months, 6 months and 12 months
  To rate satisfaction with overall teatment regime with a numerical scale of 0 (least satisfied) to 10 (most satisfied)
Pain score post-procedure | 10 days post-op
  Participants will record their pain score using the Visual Analogue Score (VAS) for pain. The scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Occulsion rates | 2-weeks, 3 months, 6 months and 12 months
  Duplex ultrasound performed at specific timepoints to ensure that the treated vein is occluded.

CONTACTS AND LOCATIONS:
Overall Officials: Tang Tjun Yip, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Background] Beebe-Dimmer JL, Pfeifer JR, Engle JS, Schottenfeld D. The epidemiology of chronic venous insufficiency and varicose veins. Ann Epidemiol. 2005 Mar;15(3):175-84. doi: 10.1016/j.annepidem.2004.05.015. PMID 15723761
- [Background] van den Bos R, Arends L, Kockaert M, Neumann M, Nijsten T. Endovenous therapies of lower extremity varicosities: a meta-analysis. J Vasc Surg. 2009 Jan;49(1):230-9. doi: 10.1016/j.jvs.2008.06.030. Epub 2008 Aug 9. PMID 18692348
- [Background] Geza M, Gloviczki P. Venous Embryology and Anatomy. In: Bergan JJ, editor. The Vein Book: Elsivier Academic Press; 2007.
- [Background] van Eekeren RR, Boersma D, de Vries JP, Zeebregts CJ, Reijnen MM. Update of endovenous treatment modalities for insufficient saphenous veins--a review of literature. Semin Vasc Surg. 2014 Jun;27(2):118-36. doi: 10.1053/j.semvascsurg.2015.02.002. Epub 2015 Feb 18. PMID 25868763
- [Background] Guex JJ. Endovenous chemical (and physical) treatments for varices: what's new? Phlebology. 2014 May;29(1 suppl):45-48. doi: 10.1177/0268355514526331. Epub 2014 May 19. PMID 24843085
- [Background] Davies HO, Popplewell M, Darvall K, Bate G, Bradbury AW. A review of randomised controlled trials comparing ultrasound-guided foam sclerotherapy with endothermal ablation for the treatment of great saphenous varicose veins. Phlebology. 2016 May;31(4):234-40. doi: 10.1177/0268355515595194. Epub 2015 Jul 9. PMID 26163507